CLINICAL TRIAL: NCT00449930
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of Sitagliptin Compared With Metformin in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control
Brief Title: Sitagliptin Comparative Study in Patients With Type 2 Diabetes (0431-049)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-049; MK0431-049; 2006_561
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug
  Interventions: Drug: sitagliptin phosphate
- 2 (Active Comparator): Active comparator
  Interventions: Drug: Comparator: metformin hydrochloride

INTERVENTIONS:
Drug: sitagliptin phosphate — (1) sitagliptin 100mg tablet once daily (q.d.) for a 24-wk treatment period
  Other Names: MK0431
  Arms: 1
Drug: Comparator: metformin hydrochloride — (4) Metformin 500mg tablets once daily (q.d.) for a 24-wk treatment period.
  Arms: 2

SUMMARY:
A study to evaluate the efficacy and safety of sitagliptin in comparison to a commonly used medication in patients with type 2 diabetes

ELIGIBILITY:
General Inclusion Criteria:

* Patient has type 2 diabetes mellitus (T2DM)
* Patient is inadequately controlled and not on treatment with insulin or oral antihyperglycemic therapy

General Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient was on antihyperglycemic therapy (insulin or oral) within the prior 4 months

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2008-07-25 (Actual); Study Completion 2008-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Aschner P, Katzeff HL, Guo H, Sunga S, Williams-Herman D, Kaufman KD, Goldstein BJ; Sitagliptin Study 049 Group. Efficacy and safety of monotherapy of sitagliptin compared with metformin in patients with type 2 diabetes. Diabetes Obes Metab. 2010 Mar;12(3):252-61. doi: 10.1111/j.1463-1326.2009.01187.x. Epub 2009 Nov 25. PMID 20070351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient In: 04-Apr-2007
  Last Patient Last Visit: 25-Jul-2008
  113 study centers worldwide
Pre-assignment Details: Patients 18-78 years of age with Type 2 diabetes mellitus (T2DM) who were not on anti-hyperglycemic agents for at least 4 months (16 weeks) and with a hemoglobin A1c (HbA1c) of ≥ 6.5 and ≤9.0%
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablet of sitagliptin once daily.
- Metformin: The Metformin group includes data from patients randomized to receive treatment with metformin initiated at a dose of 1 tablet (500 mg) per day. Patients were then to be up-titrated over a maximum of 5 weeks to a total daily dose of 2 tablets twice daily (1000 mg b.i.d).
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Metformin
Started | 528 | 522
Completed | 467 | 447
Not Completed | 61 | 75
Not completed — Adverse Event | 9 | 19
Not completed — Trial Terminated ( Site Closed) | 1 | 0
Not completed — Lack of Efficacy | 10 | 1
Not completed — Lost to Follow-up | 9 | 14
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 14 | 15
Not completed — Withdrawal by Subject | 16 | 23
Not completed — Glycemic discontinuation criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Metformin | Total
Number analyzed (Participants) | 528 | 522 | 1050
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.7) | 56.1 (10.4) | 56.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 288 | 566
  Male | 250 | 234 | 484
Race/Ethnicity, Customized [Number; unit: participants]
  White | 397 | 395 | 792
  Black | 24 | 19 | 43
  Asian | 64 | 62 | 126
  Other | 43 | 46 | 89
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 84.9 (17.7) | 84.6 (17.2) | 84.7 (17.5)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.2 (0.7) | 7.3 (0.7) | 7.3 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and 24 weeks
Population: The per protocol population required that a patient had measurements both at baseline and at Week 24, and did not have any major protocol violations (e.g. drug compliance <85%, addition of prohibited antihyperglycemic agent, incorrect double-blind study medication). No missing data were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Metformin
Number analyzed (Participants) | 455 | 439
Percent | -0.43 [-0.48 to -0.38] | -0.57 [-0.62 to -0.51]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Metformin; Test type: Non-Inferiority or Equivalence — The pre-specified non-inferiority margin was 0.4%; i.e., non-inferiority required that the upper boundary of the 95% confidence interval for the treatment difference (sitagliptin minus metformin) to be less than 0.4%; Mean Difference (Net) = 0.14, 95% CI [0.06 to 0.21], Standard Deviation 0.57 — Based on an analysis of covariance (ANCOVA) model with terms for treatment group and baseline value

2. Secondary Outcome: Number of Patients Who Reported 1 or More Episodes of the Adverse Experience of Diarrhea
Time Frame: Baseline to Week 24
Population: All randomized patients who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Metformin
Number analyzed (Participants) | 528 | 522
Participants
  Patients Who Reported Diarrhea | 19 | 57
  Patients Who Did Not Report Diarrhea | 509 | 465
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Metformin; Test type: Superiority or Other; p < 0.001, Fisher Exact; Risk Difference (RD) = -7.3, 95% CI [-10.6 to -4.2] — Difference (sitagliptin minus metformin) in the percentage of patients with diarrhea. Wilson Score method was used for the 95% Confidence Interval (CI)

3. Secondary Outcome: Number of Patients Who Reported 1 or More Episodes of the Adverse Experience of Nausea
Time Frame: Baseline to Week 24
Population: All randomized patients who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Metformin
Number analyzed (Participants) | 528 | 522
Participants
  Patients Who Reported Nausea | 6 | 16
  Patients Who Did Not Report Nausea | 522 | 506
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Metformin; Test type: Superiority or Other; p = 0.032, Fisher Exact; Risk Difference (RD) = -1.9, 95% CI [-3.9 to -0.2] — Difference (sitagliptin minus metformin) in the percentage of patients with nausea. Wilson Score method was used for the 95% CI

4. Secondary Outcome: Number of Patients Who Reported 1 or More Episodes of the Adverse Experience of Abdominal Pain
Time Frame: Baseline to Week 24
Population: All randomized patients who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Metformin
Number analyzed (Participants) | 528 | 522
Participants
  Patients Who Reported Abdominal Pain | 11 | 20
  Patients Who Did Not Report Abdominal Pain | 517 | 502
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Metformin; Test type: Superiority or Other; p = 0.103, Fisher Exact; Risk Difference (RD) = -1.7, 95% CI [-4.0 to 0.3] — Difference (sitagliptin minus metformin) in the percentage of patients with abdominal pain. Wilson Score method was used for the 95% CI

5. Secondary Outcome: Number of Patients Who Reported 1 or More Episodes of the Adverse Experience of Vomiting
Time Frame: Baseline to Week 24
Population: All randomized patients who received at least 1 dose of the double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg | Metformin
Number analyzed (Participants) | 528 | 522
Participants
  Patients Who Reported Vomiting | 2 | 7
  Patients Who Did Not Report Vomiting | 526 | 515
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Metformin; Test type: Superiority or Other; Risk Difference (RD) = -1.0, 95% CI [-2.4 to 0.2] — Difference (sitagliptin minus metformin) in the percentage of patients with vomiting. Wilson Score method was used for the 95% CI

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg | Metformin
Serious Adverse Events (participants affected / at risk) | 10 | 8
Other Adverse Events (participants affected / at risk) | 19 | 57
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg | Metformin
Any Cardiac disorders (Cardiac disorders) | 1/528 | 3/522
Acute myocardial infarction (Cardiac disorders) | 0/528 | 1/522
Angina pectoris (Cardiac disorders) | 1/528 | 0/522
Coronary artery disease (Cardiac disorders) | 0/528 | 1/522
Tachyarrhythmia (Cardiac disorders) | 0/528 | 1/522
Any Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0/528 | 1/522
Multiple endocrine adenomatosis Type II (Congenital, familial and genetic disorders) | 0/528 | 1/522
Any General disorders and administration site conditions (General disorders) | 0/528 | 1/522
Non-cardiac chest pain (General disorders) | 0/528 | 1/522
Any Infections and infestations (Infections and infestations) | 2/528 | 2/522
Appendicitis (Infections and infestations) | 1/528 | 0/522
Cellulitis (Infections and infestations) | 0/528 | 1/522
Gastroenteritis (Infections and infestations) | 1/528 | 0/522
Upper respiratory tract infection (Infections and infestations) | 0/528 | 1/522
Any Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3/528 | 0/522
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1/528 | 0/522
Joint injury (Injury, poisoning and procedural complications) | 1/528 | 0/522
Tibia fracture (Injury, poisoning and procedural complications) | 1/528 | 0/522
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1/528 | 0/522
Hypoglycaemia (Metabolism and nutrition disorders) | 1/528 | 0/522
Any Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/528 | 1/522
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/528 | 0/522
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/528 | 1/522
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/528 | 0/522
Any Nervous system disorders (Nervous system disorders) | 1/528 | 0/522
Facial palsy (Nervous system disorders) | 1/528 | 0/522
Any Renal and urinary disorders (Renal and urinary disorders) | 1/528 | 0/522
Nephrolithiasis (Renal and urinary disorders) | 1/528 | 0/522
Any Reproductive system and breast disorders (Reproductive system and breast disorders) | 0/528 | 1/522
Hydrometra (Reproductive system and breast disorders) | 0/528 | 1/522
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg | Metformin
Any Gastrointestinal disorders (Gastrointestinal disorders) | 19/528 | 57/522
Diarrhoea (Gastrointestinal disorders) | 19/528 | 57/522

LIMITATIONS AND CAVEATS:
Site 0490125 was non-compliant with Good Clinical Practice (GCP). Data from the 8 patients at this site were removed from all analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.